CLINICAL TRIAL: NCT07024134
Title: Recovery Optimization: Adding Tissue Flossing to Nerve Glide on Axillary Web Syndrome Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005818
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Axillary Web Syndrome
Keywords: mastectomy; nerve glide; tissue flossing

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Shoulder flossing with ROM exercises (Experimental)
  Interventions: Other: Shoulder flossing application
- Nerve Glide exercises (Experimental)
  Interventions: Other: Nerve glide application
- Shoulder flossing with Nerve Glide (Experimental)
  Interventions: Other: Shoulder flossing with Nerve Glide
- Control group (No Intervention)

INTERVENTIONS:
Other: Shoulder flossing application — Select a floss band, typically made of latex, which is about 1-2 inches wide. Ensure the area to be wrapped is clean and dry to prevent slipping. Begin wrapping the floss band around the upper arm, just below the shoulder joint. Start at the deltoid's base. Leave about 2 inches of the band free at the start to tuck in the end when you finish wrapping. Wrap the band tightly but not to the point of causing discomfort or cutting off circulation, the band should be snug but not so tight that it causes numbness or tingling. Aim for about a 50% stretch of the band as you wrap. Continue wrapping down the arm, covering the entire upper arm and ending just above the elbow Overlap each layer by about 50% to ensure even coverage and compression. Once you reach the desired coverage area, tuck the end of the band under the last loop to secure it. Check the tightness to ensure it is snug but not overly constrictive.
  Arms: Shoulder flossing with ROM exercises
Other: Nerve glide application — With the band in place, perform slow and controlled arm movements. Start with shoulder abduction (lifting the arm sideways) and progress to external rotation (turning the arm outward) this is for axillary nerve glide, (extending your arm and fingers while tilting your head away from the affected side) this for median nerve glide and (Extend your arm out to the side at shoulder height-Rotate the arm so the palm faces upwards-Flex the wrist and fingers back gently-Tilt your head away from the extended arm to increase the stretch) this for radial nerve glide. Ensure movements are within a pain-free range. Stop if any discomfort occurs. Keep the floss band in place for 1-2 minutes while performing nerve glides. Remove the band after the exercise, allowing the skin to recover from compression.
  Arms: Nerve Glide exercises
Other: Shoulder flossing with Nerve Glide — Procedures of Shoulder flossing application adding to Procedures of Nerve glide application.
  Arms: Shoulder flossing with Nerve Glide

SUMMARY:
Axillary web syndrome (AWS) is a complication associated with breast cancer surgery, characterized by pain, functional limitation of the shoulder and decreased quality of life. There are several physical treatment options to reduce pain and improve the functionality of the upper limb in women with AWS. This study evaluates the effectiveness of an early rehabilitation approach to prevent axillary web syndrome consisting in functional and proprioceptive re-education, manual lymphatic drainage and kinesio taping after breast cancer surgery.

DETAILED DESCRIPTION:
Tissue flossing for the upper limb involves wrapping a floss band, typically made of elastic material, around the targeted area to provide compression and create a shearing effect on the tissue. This technique is utilized to enhance mobility, reduce pain, and improve recovery. The procedure begins by wrapping the band around the upper limb, starting from the distal part of the limb and moving proximally, ensuring a snug but not overly tight application that allows for some movement. The band is usually left in place for approximately 2-3 minutes. Physiologically, Tissue flossing for the upper limb, often referred to as compression wrapping, plays a significant role in enhancing physiological functions by improving joint mobility and reducing pain. This technique involves tightly wrapping a stretchable band around a muscle or joint to create compression. The compression temporarily restricts blood flow, which, upon release, results in a rush of blood back to the tissues. This process enhances circulation, promoting nutrient delivery and waste removal from the affected area.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 45 and 65 years with diagnosis of breast cancer underwent to quadrantectomy and axillary lymphadenectomy.
* No change of arm size.
* Females only will participate in the study.
* All patients have axillary web syndrome
* All patients' relatives enrolled to the study will have their informed consent

Exclusion Criteria:

* Metastatic disease, infections, past TVP, emboli.
* Lymphedema.
* Chemotherapy and Radiotherapy.
* Pregnant women.
* Patients who suffer from mental or psychological problems.
* Patients who have psoriasis, liver disease, diabetes mellitus, hypertensive patients and cardiac -robleme
* Patients have Genetic disease or deformity
* Who has previous injury or fracture in shoulder joint
* Rheumatoid arthritis
* Osteopenia
* Frozen shoulder
* metastases of any kind
* lymphedema,
* a traumatic injury to the targeted upper extremity
* a musculoskeletal disorder
* taking any anticoagulants
* had undergone bilateral breast cancer surgery
* experienced locoregional recurrence
* had vascular problems in the affected upper extremity

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female with post mastectomy axillary web syndrome
Enrollment: 155 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain. Visual Analogic Scale (VAS): | at baseline and at 12 weeks
  According to the National Cancer Institute (NIH), it is a tool used to help the professional assess the intensity of certain sensations and feelings, such as pain. The Visual Analog Scale in Arabic version for pain is composed of a straight line on which an extreme means no pain and the other extreme means the worst pain imaginable.
axillary cord thickness | at baseline and at 12 weeks
  Ultrasonography, this device will be used for the assessment of axillary cord thickness, echogenicity and disorganization. One technique used in ultrasonography is utilizing a high-resolution ultrasound system with 18 MHz frequency, which provides high-definition superficial imaging. A gel technique is also used to reduce artifacts caused by tissue compression. This technique can be used to measure cord thickness, echogenicity, and disorganization.

SECONDARY OUTCOMES:
Shoulder Range of Movement (flexion, extension, abduction and external and internal rotation) | at baseline and at 12 weeks
  The investigators will use Goniometry of affected shoulder .The patients were asked to move their arms in flexion, extension, abduction and external and internal rotation of the shoulder.
Quality of life. Barthel Scale: | at baseline and at 12 weeks
  The Barthel index or Barthel scale is an instrument used in Arabic version by social and health professionals for the functional assessment of a patient and to monitor their evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No